CLINICAL TRIAL: NCT04006093
Title: Pharmacokinetics of Apixaban in Subjects With End-stage Renal Disease Treated With Peritoneal Dialysis: the ApiDP Study
Brief Title: Apixaban in Subjects With Peritoneal Dialysis
Acronym: ApiDP
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Hospital, Caen (Other)
Collaborators: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 19-060
Record Dates: First submitted 2019-06-05; First posted 2019-07-02 (Actual); Last update posted 2023-01-20 (Actual); Status verified 2019-04

CONDITIONS: Chronic Renal Insufficiency; Peritoneal Dialysis
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — apixaban

STUDY DESIGN:
Intervention Model Description: Two groups of participants will receive one single-dose of 5 mg of apixaban: the first group of participants with a normal renal function, the second group contains participants with end-stage renal disease treated with peritoneal dialysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- participants with normal renal function (Experimental)
  Interventions: Drug: Apixaban Oral
- participants with end-stage renal disease (Experimental)
  Interventions: Drug: Apixaban Oral

INTERVENTIONS:
Drug: Apixaban Oral — one Tablet 5mg

SUMMARY:
The primary objective of this study is to assess the pharmacokinetics of a single oral dose of apixaban (5mg) in participants with dialysis peritoneal versus participants with normal renal function.

DETAILED DESCRIPTION:
Participants with chronic renal disease treated with peritoneal dialysis and participants with normal renal function are hospitalized for three days.

ELIGIBILITY:
Inclusion Criteria:

* Participant with 21<BMI<40
* French participant
* Participant able to consent
* Participant with social insurance
* Participant on peritoneal dialysis for at least 3 months with end-stage renal disease treated

Exclusion Criteria:

* Participant with hypersensibility reactions to apixaban
* Participant with a history of major bleeding
* Participant already on anticoagulant
* Participant on non-stearoid anti-inflammatory at anti-inflammatory dosage > 300 mg
* Participant on potent inhibitors of CYP 3A4 and P-gp
* Participant on inducers of CYP3A4 and P-sp
* Participant with moderate (Child-Pugh B) or severe (Child-Pugh C) hepatic impairment
* Participant receiving or having received antibiotic treatment within 14 days prior to study
* Pregnant or lactating women
* Participant with known hypersensitivity reactions to icodextrin
* Participant not supporting an intraperitoneal volume of 2 liters (only participant with peritoneal dialysis)
* Participant with "Normal renal function" with glomerular filtration rate < 90 ml/min

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2019-12-08 (Actual); Primary Completion 2022-12-10 (Actual); Study Completion 2022-12-10 (Actual)

PRIMARY OUTCOMES:
Apixaban area Under the curve | Day 3
  Measurement of apixaban plasma concentrations at different times.
Apixaban maximum plasma concentration | Day 3
  Measurement of apixaban plasma concentrations at different times.

SECONDARY OUTCOMES:
anti-Xa activity | Hour 0, Hour 3, Hour 9 and Hour 72
  anti-Xa activity plasma measurements
TP activity | Hour 0, Hour 3, Hour 9 and Hour 72
  TP activity plasma measurements
TCA activity | Hour 0, Hour 3, Hour 9 and Hour 72
  TCA activity plasma measurements
Apixaban urinary elimination | Day 3
  Measurement of apixaban urinary concentrations
Apixaban maximum peritoneal concentration | day 3
  Measurement of apixaban peritoneal fluid concentrations

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Caen, Caen, France

IPD SHARING:
Plan to Share IPD: Undecided